CLINICAL TRIAL: NCT01874574
Title: Intra-articular Corticosteroid Injection Compared With Single-Shot Hyaluronic Acid for Treatment of Osteoarthritis Knee: A Prospective, Double-blind Randomized Controlled Trial
Brief Title: Intra-articular Corticosteroid Injection Compared With Single-Shot Hyaluronic Acid for Treatment of Osteoarthritis Knee
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Phonthakorn Panichkul, Dr. Phonthakorn Panichkul, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OrthoTU-01
Record Dates: First submitted 2012-09-05; First posted 2013-06-11 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Corticosteroid; Hyaluronic acid; Intra-articular injection
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — hylan; Adrenal Cortex Hormones; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single shot Hylan G-F 20 (Synvisc) (Experimental): Intra-articular injection of the Single shot 6 mL of Hylan G-F 20 (Synvisc)
  Interventions: Drug: Hylan G-F 20
- Corticosteroid (Triamcinolone acetonide) (Active Comparator): Intra-articular injection of 1 mL of 40 mg Triamcinolone acetonide plus 5 mL of 1% xylocaine with adrenaline injected at the knee by single shot
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Drug: Hylan G-F 20 — After full aseptic preparation, Single shot intra-articular injection either 6 mL of Hylan G-F 20 or 1 mL of 40 mg triamcinolone acetonide plus 5 mL of 1% xylocaine with adrenaline were injected into the joint cavity using the infero-lateral approach via a 21-gauge needle.
  Other Names: Synvisc
  Arms: Single shot Hylan G-F 20 (Synvisc)
Drug: Corticosteroid — After full aseptic preparation, Single shot intra-articular injection either 6 mL of Hylan G-F 20 or 1 mL of 40 mg triamcinolone acetonide plus 5 mL of 1% xylocaine with adrenaline were injected into the joint cavity using the infero-lateral approach via a 21-gauge needle.
  Other Names: Triamcinolone acetonide
  Arms: Corticosteroid (Triamcinolone acetonide)

SUMMARY:
Corticosteroid and Hylan G-F 20 are both effective in improving pain and function of osteoarthritic knee patients.

DETAILED DESCRIPTION:
Corticosteroid and Hylan G-F 20 are both effective in improving pain and function of osteoarthritic knee patients up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of knee OA
* Knee pain for most days of the prior month
* Radiographic evidence consistent with knee OA
* Aged between 40 and 80 years old

Exclusion Criteria:

* Lumbar spondylosis
* Gross deformity of the knee
* Co-existent inflammatory or crystal arthritis
* Prior knee surgery
* Injury to the knee in the preceding 6 months
* Any intra-articular injection in the preceding 3 months
* Pregnant or Lactating
* Current infection in the affected knee
* Inability to provide informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
WOMAC Score | 6 months
  Change from Baseline in WOMAC score at 6 months

SECONDARY OUTCOMES:
Visual Analogue Scale(VAS) | 6 months
  Change from Baseline in VAS score at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nattapol Tammachote, MD, MSc, Study Director — Department of Orthopaedics, Thammasat University
Locations (1):
- Thammasat University Hospital, Thammasat University, Prathumthani, Changwat Pathum Thani, Thailand